CLINICAL TRIAL: NCT06052800
Title: An Observational Study of Enzyme Replacement Therapy-Naïve and Agalsidase Beta-Treated Fabry Disease Patients With GLA IVS4 919 G>A Mutation in Taiwan
Brief Title: Agalsidase Beta Long-Term Treatment Outcome for Fabry Disease Patients With IVS4 Mutation in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17349; U1111-1287-7177 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Patients with Galactosidase Alpha gene (GLA) IVS4 who have already received agalsidase beta treatment
- Cohort 2: Patients with GLA IVS4 who will initiate agalsidase beta treatment
- Cohort 3: Enzyme replacement therapy (ERT)-naive Fabry disease patients with GLA IVS4

SUMMARY:
This is a national, multicenter, observational, cohort study designed to assess clinical outcomes upon agalsidase beta treatment, to characterize the clinical manifestations, and to collect the natural history on male and female Fabry disease adult patients who carry the GLA IVS4.

This study aims to retrospectively and prospectively investigate the disease natural history, clinical manifestations, and the treatment outcomes upon agalsidase beta in Fabry disease (FD) patients carrying the GLA IVS4 mutation from medical records, physician assessments, and patient-reported outcomes.

DETAILED DESCRIPTION:
Study Design Time Perspective: Retrospective and Prospective

ELIGIBILITY:
Inclusion Criteria:

- Provide signed informed consent.

Cohort 1:

* Male or female Fabry disease patient with documented GLA IVS4 in medical record.
* Age ≥ 18 years old at the time of signing informed consent.
* The maximum proportion of female is 20% of cohort 1.
* Patient who has received agalsidase beta treatment for at least 6 months.
* The data of LVMI, LPWT, IVST and blood lyso-Gb3 concentration are all available within 6 months prior to agalsidase beta treatment initiation.

Cohort 2:

* Male or female Fabry disease patient with documented GLA IVS4 in medical record.
* Age ≥ 18 years old at the time of signing informed consent.
* The maximum proportion of female is 20% of cohort 2.
* Patient who plans to apply for the National Health Insurance Reimbursement for agalsidase beta medication.
* The data of LVMI, LPWT, IVST and blood lyso-Gb3 concentration are all available within 6 months prior to agalsidase beta treatment initiation.

Cohort 3:

* Male or female Fabry disease patients with documented GLA IVS4 mutation in medical record.
* Male patient is aged ≥ 30 years old and female patient is aged ≥ 40 years old at the time of signing informed consent.
* The maximum proportion of female is 20% of cohort 3.
* Patient who has never received agalsidase alpha or agalsidase beta treatment (ERT-naïve).
* Elevated blood lyso-Gb3.
* At least ONE of the following conditions documented in medical record:

  1. cardiac parameter abnormalities (e.g. via imaging, electrophysiology, or biomarker);
  2. at least one FD-related sign/symptom.
* The data of LVMI, LPWT, IVST and blood lyso-Gb3 concentration are all available within 6 months.
* Patients who are expected not to receive ERT or FD-specific treatment per investigator's judgement.

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, may interfere with patient's participation in the study, such as life expectancy of less than 6 months (e.g. diagnosed with malignancy, CAD)
* Fabry patients who have severe heart disease (NYHA Class IV) or severe myocardial fibrosis per investigator judgement
* Known non-Fabry disease infiltrative cardiomyopathy including amyloidosis
* Known non-GLA genetic (e.g., sarcomeric, metabolic mutations) hypertrophic cardiomyopathy.
* Patients who are receiving any Fabry disease-specific treatment (enzyme replacement therapy, chaperone therapy, substrate reduction therapy, or gene therapy) other than agalsidase beta for Fabry disease
* Pregnancy or suspected pregnancy
* Patient diagnosed with moderate to severe dementia
* Unstable patient condition as judged by investigator (e.g., hypertension, diabetes, and systematic disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FD patients carrying the GLA IVS4 mutation, who are eligible for 1 of the cohorts (1, 2, 3).
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: change of Left ventricular mass index (LVMI) as measured by echocardiography in agalsidase beta-treated patients | through study completion with a minimum of 2 years
Cohort 2: change of Left ventricular mass index (LVMI) as measured by echocardiography in agalsidase beta-treated patients | up to 1.5 years

SECONDARY OUTCOMES:
Change of Left posterior wall thickness (LPWT) as measured by echocardiography | For cohort 1, through study completion with a minimum of 2 years For cohort 2, 1.5 years For cohort 3, through study completion with a minimum of 1.5 years
Change of Interventricular septal thickness (IVST) as measured by echocardiography | For cohort 1, through study completion with a minimum of 2 years For cohort 2, 1.5 years For cohort 3, through study completion with a minimum of 1.5 years
Change of blood Globotriaosylsphingosine (lyso-Gb3) concentration | For cohort 1, through study completion with a minimum of 2 years For cohort 2, 1.5 years For cohort 3, through study completion with a minimum of 1.5 years
Change of left ventricular mass index (LVMI) as measured by echocardiography in ERT-naive patients | For cohort 3, through study completion with a minimum of 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (5):
- Taiwan (5):
  - Investigational Site Number : 1580004, Taichung
  - Investigational Site Number : 1580005, Tainan
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1580002, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org